CLINICAL TRIAL: NCT03245944
Title: Optimal Timing of Percutaneous Intervention in Non-maturing Dialysis Fistulas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Alian Al-Balas, Prinicipal investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F0001
Record Dates: First submitted 2017-07-31; First posted 2017-08-10 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Immature Arteriovenous Fistula
Keywords: immature AVF; percutaneous intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- early angioplasty (Active Comparator): Patients who initiated hemodialysis with a CVC, then had a new AVF created after commencing dialysis, and then had a 6-week postoperative ultrasound that revealed an immature AVF (diameter < 4 mm diameter or blood flow < 500 ml/min). These patients who an early angioplasty intervention group that will undergo a routine Angioplasty at 6 weeks after AVF creation
  Interventions: Procedure: early Angioplasty
- late Angioplasty (Experimental): Patients who initiated hemodialysis with a CVC, then had a new AVF created after commencing dialysis, and then had a 6-week postoperative ultrasound that revealed an immature AVF (diameter < 4 mm diameter or blood flow < 500 ml/min). These patients who a late angioplasty intervention group in which early Angioplasty will be avoided and subsequently be performed only if the 3-month ultrasound indicates persistent AVF immaturity
  Interventions: Procedure: late Angioplasty

INTERVENTIONS:
Procedure: early Angioplasty — Angioplasty is a minimally invasive, endovascular procedure to widen narrowed or obstructed arteries or veins. A deflated balloon attached to a catheter (a balloon catheter) is passed over a guide-wire into the narrowed vessel and then inflated to a fixed size. The balloon forces expansion of the blood vessel and the surrounding muscular wall, allowing an improved blood flow. This is part of standard of care for immature arteriovenous fistulas. Early means pt will get the procedure at 6 weeks from time of initiation of AVFs
  Other Names: Early PTA
  Arms: early angioplasty
Procedure: late Angioplasty — Angioplasty is a minimally invasive, endovascular procedure to widen narrowed or obstructed arteries or veins. A deflated balloon attached to a catheter (a balloon catheter) is passed over a guide-wire into the narrowed vessel and then inflated to a fixed size. The balloon forces expansion of the blood vessel and the surrounding muscular wall, allowing an improved blood flow. This is part of standard of care for immature arteriovenous fistulas. Late means the angioplasty is done at 3 months from time of AVF creation if still immature at that time.
  Other Names: Late PTA
  Arms: late Angioplasty

SUMMARY:
Arteriovenous fistulas (AVFs) are the preferred type of vascular access for dialysis, but many of them fail to mature. The optimal timing of intervention to salvage immature AVFs is unknown.The study proposes a randomized clinical trial comparing the clinical and economic impact of early vs late angioplasty in non-maturing AVFs.

The study proposes a RCT to test the hypothesis that, as compared to early angioplasty of non-maturing AVFs, late angioplasty results in a lower proportion of AVFs being used at 6 months, but a greater long-term AVF patency , lower requirement of subsequent interventions to maintain AVF patency for dialysis, and lower overall cost of access maintenance.

DETAILED DESCRIPTION:
The optimal timing of intervention in non-maturing AVFs remains controversial, and can only be definitively addressed by a randomized clinical trial (RCT) comparing early (6 weeks) vs late (3 months) angioplasty of non-maturing AVFs. The investigators will perform a single-center, prospective RCT. The investigators will recruit 112 patients who initiated hemodialysis with a CVC, then had a new AVF created after commencing dialysis, and then had a 6-week postoperative ultrasound that revealed an immature AVF (diameter < 4 mm diameter or blood flow < 500 ml/min). These patients will be randomized to one of two groups: an early intervention group that will undergo a routine PTA at 6 weeks after AVF creation, or a late intervention group in which early PTA will be avoided and subsequently be performed only if the 3-month ultrasound indicates persistent AVF immaturity. These patients will be followed for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with End stage renal disease (ESRD).
* Patients on hemodialysis.
* Patients using central venous catheter (CVC).
* Patients who had a new AVF created after commencing dialysis.
* Patients who had immature fistula ( 6-week postoperative ultrasound that revealed an immature AVF (diameter < 4 mm diameter or blood flow < 500 ml/min).

Exclusion Criteria:

• Children with Age below 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Fistula Maturity | baseline- 6 months
  Ultrasound of the fistula:
  Mature fistula Criteria:
  1. Blood flow of at least 500 ml/min and
  2. Minimum diameter of 4 mm

SECONDARY OUTCOMES:
Fistula survival | baseline-2 years
  Ultrasound of the fistula:
  1. Blood flow of at least 500 ml/min and
  2. Minimum diameter of 4 mm
Fistula adequacy | Baseline- 2 years
  Fistula is used for hemodilaysis and provide adequate clearance which is measured by:
  Kt/V: 1.4 where K: clearance [m3/s], t: time [m3/s], V:volume of distribution [m3]

CONTACTS AND LOCATIONS:
Locations (1):
- UAB, Birmingham, Alabama, United States

REFERENCES:
- [Background] Al-Balas A, Lee T, Young CJ, Barker-Finkel J, Allon M. Predictors of Initiation for Predialysis Arteriovenous Fistula. Clin J Am Soc Nephrol. 2016 Oct 7;11(10):1802-1808. doi: 10.2215/CJN.00700116. Epub 2016 Sep 14. PMID 27630181
- [Background] Al-Balas A, Lee T, Young CJ, Kepes JA, Barker-Finkel J, Allon M. The Clinical and Economic Effect of Vascular Access Selection in Patients Initiating Hemodialysis with a Catheter. J Am Soc Nephrol. 2017 Dec;28(12):3679-3687. doi: 10.1681/ASN.2016060707. Epub 2017 Jul 14. PMID 28710090